CLINICAL TRIAL: NCT02563938
Title: A Phase 1, Randomized, Double-Blind, Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AK001 in Subjects With Atopic Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AK001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK001-001
Record Dates: First submitted 2015-09-15; First posted 2015-09-30 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Atopy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AK001 (Experimental): Up to six single ascending doses of AK001.
  Interventions: Drug: AK001
- Saline Solution (Placebo Comparator): Saline solution will be administered as a single infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK001 — Given parenterally.
  Arms: AK001
Drug: Placebo
  Other Names: Saline solution
  Arms: Saline Solution

SUMMARY:
This first-in-human study will evaluate the safety and tolerability of single doses of AK001 across a range of potentially active doses. Early signals of pharmacodynamic activity will also be evaluated.

DETAILED DESCRIPTION:
AK001 is a monoclonal antibody which may be useful in the treatment of patients with severe allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-30
* Determined to be in good health
* Clinical laboratory values within limits of normal values
* Normal 12-lead ECG
* Stool sample negative for parasites
* Non-smoker
* Consumed an average of no more than 2 drinks per day within 6 months
* Subjects of reproductive age must use a highly effective method of contraception
* Positive skin test in certain cohorts
* Elevated total eosinophil counts in certain cohorts

Exclusion Criteria:

* Clinically significant medical history conditions or laboratory values
* Receipt of investigational drug, biologic or medical device within 30 days prior to Screening
* New drug therapy within 1 week of study drug administration
* Antihistamine use within 2 weeks prior to Screening
* Consumption of alcohol within 48 hours of study drug administration
* Positive urine drug test or cotinine test at Screening or Day -1
* History, within the last 2 years, of alcohol abuse, illicit drug use, or significant mental illness
* Demonstration of veins unsuitable for repeated venipuncture or IV infusion
* Recent treatment with alternative therapies which may confound clinical or laboratory assessments
* Donation or loss of more than 500 mL of blood within 56 days prior to study drug administration
* History of malignancy within last 5 years
* History of severe allergic or anaphylactic reactions
* Females who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of AK001 measured by number of subjects with adverse events and dose limiting toxicities (DLTs) respectively | Within 86 days

SECONDARY OUTCOMES:
Immediate hypersensitivity skin testing | Within 28 days
Peripheral blood counts for eosinophils and basophils | Within 28 days
Serum eosinophilic cationic protein (ECP) and tryptase levels | Within 28 days
24-hour urine measurement of histamine, N-methylhistamine, and 11-beta-prostaglandin F2 | Within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — Allakos Inc.
Locations (1):
- Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided